CLINICAL TRIAL: NCT01757314
Title: A Prospective Study Comparing Palpation Guided and Ultrasound Guided Arterial Catheter Placement by Anesthesiology Residents in Training
Brief Title: Comparing Palpation Guided and Ultrasound Guided Arterial Line Placement
Status: Terminated | Type: Observational
Why Stopped: already several publications in the literature
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Sponsor
Other Study IDs: 2012001193
Record Dates: First submitted 2012-09-27; First posted 2012-12-28 (Estimated); Last update posted 2016-09-28 (Estimated); Status verified 2015-09

CONDITIONS: Surgeries Requiring Arterial Lines
Keywords: arterial lines
MeSH Terms: interventions — High-Energy Shock Waves

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- CA 1 and 2 anethesia residents: palpation technique
  Interventions: Other: palpation technique
- Ca1 and 2 residents: ultrasound guided technique
  Interventions: Behavioral: ultrasound technique

INTERVENTIONS:
Behavioral: ultrasound technique — instruction in the ultrasound technique
  Groups: Ca1 and 2 residents
Other: palpation technique — placement of a line via palpation technique
  Groups: CA 1 and 2 anethesia residents

SUMMARY:
When surgery is performed under general anesthesia, a catheter is placed in a vein to administer drugs and saline. During major operations, an additional catheter is placed in an artery in order to measure the blood pressure closely and withdraw blood samples at frequent intervals for various laboratory tests. This arterial catheter is usually placed by feeling the patient's artery at the wrist and inserting the guide-needle in a blind fashion. This procedure, at times, leads to delays and failures due to an inability to feel the arterial pulsation well either due to the patients' anatomy or the anesthetic effect. This study will determine whether training Anesthesiology Residents in the use of ultrasound technology and its application in identifying an artery can prevent the problems associated with the conventional palpation technique. Our finding will lead to better and safer anesthetic management of patients presenting for a major surgical procedure. Furthermore, the finding will help us in introducing the education and training of ultrasound-guided arterial catheter placement in our Residency Program.

The investigators propose to follow anesthesia residents over a course of 3 years assessing their skill level for both palpation and ultrasound technique.

DETAILED DESCRIPTION:
This is an updated study on a previous IRB-approved research (0120070296) which was terminated prior to conclusion as the principal investigator terminated his employment at the UNDNJ. An arterial catheter is routinely placed immediately following induction of anesthesia, in major operative procedures, in order to measure blood pressure continuously, perform frequent blood-gas analysis and withdraw blood for repeated laboratory testing. The arterial catheter is traditionally placed blindly by palpating the radial artery of the patient. This way of placing a radial artery catheter can encounter delay or failure due to conditions such as obesity, arteriosclerosis, arterial spasm and anesthesia-induced hypotension. Our study will compare the performance of Anesthesiology Residents in placing an arterial catheter by the traditional palpation-guided technique and by the ultrasound-guided technique after training in ultrasound usage. The comparison will utilize the following parameters:

* Time taken to successfully place a catheter
* Number of attempts needed to place a catheter
* Number of puncture site changes encountered
* Failure rate of the resident with each technique
* The need for replacement of the catheter during surgery The data collection will be done by an independent observer, who is not a member of the anesthesia care team or research team. The Residents performing the catheter placement will not be members of the research team and will not have access to the data. If the Resident fails to place the catheter, the attending anesthesiologist will rescue by placing the arterial catheter himself by a method of his choice. In the previous study, there was a trend toward a reduced failure rate and a decreased time for insertion with the ultrasound technique. In this study, the investigators will introduce the research to the first-year Residents and repeat the exercise during their second and third year of training in a longitudinal fashion to assess the progress during anesthesia training. The investigators plan to enroll eight residents from the first-year class. Each resident will perform eight arterial catheter placements with each technique. In addition, compared to the previous study, a more advanced ultrasound machine will be used which will provide better visualization of the radial artery.

ELIGIBILITY:
Inclusion Criteria:

* resident in training is agreeable to consent

Exclusion Criteria:

* None

Ages: 25 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: CA 1 and CA 2 residents assigned to surgical patients who require arterial lines due to complex surgical procedures
Sampling Method: Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2012-10; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
time to successful placement of catheter | residents to be timed over 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital, Newark, New Jersey, United States